CLINICAL TRIAL: NCT07329686
Title: Clinical Study of Intrastromal Anti-VEGF Injection for Corneal Neovascularization.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0998
Record Dates: First submitted 2025-12-07; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-10

CONDITIONS: Herpes Simplex Keratitis; Corneal Neovascularization
Keywords: Herpes Simplex Keratitis; corneal neovascularization
MeSH Terms: conditions — Keratitis, Herpetic; Corneal Neovascularization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group received intrastromal corneal injections of anti-VEGF (Vascular Endothelial Growth Factor) medication in conjunction with antiviral medication therapy.
  Interventions: Drug: Intrastromal anti-VEGF injection and topical antiviral eye drops
- Control group (Active Comparator): The control group was treated with conventional antiviral topical ocular drops.
  Interventions: Drug: Conventional antiviral topical ocular drops.

INTERVENTIONS:
Drug: Intrastromal anti-VEGF injection and topical antiviral eye drops — The experimental group received intrastromal corneal injections of anti-VEGF (Vascular Endothelial Growth Factor) medication in conjunction with antiviral medication therapy
  Arms: Experimental group
Drug: Conventional antiviral topical ocular drops. — The control group was treated with conventional antiviral topical ocular drops.
  Arms: Control group

SUMMARY:
Corneal stromal injection is an emerging local drug delivery method, characterized by strong targeting, high drug concentration, and prolonged duration of action. It has been preliminarily applied in the treatment of fungal keratitis and neurotrophic corneal diseases. This study aims to investigate the safety and efficacy of anti-VEGF drugs delivered via corneal stromal injection in neovascularization caused by HSK (Herpes Simplex Keratitis). The study has clear medical significance and technical feasibility, and it is expected to promote innovation in the treatment paradigm for corneal neovascularization.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Patients who meet the diagnostic criteria for Herpes Simplex Virus (HSV) keratitis with neovascularization.
* Age: Adults aged 18 years or older.
* Previous Treatment: Patients who have not undergone other anti-VEGF treatments or corneal surgeries.
* Informed Consent: Patients who are capable of understanding and signing an informed consent form, agreeing to participate in the entire study process and to follow the study's follow-up schedule and treatment plan.
* Other: Additional criteria as deemed necessary by the investigator.

Exclusion Criteria:

* Risk of Corneal Perforation: Patients at risk of corneal perforation.
* Severe Ocular Surface Dryness: Patients with severe dry eye syndrome.
* Systemic Diseases: Patients with systemic diseases that may affect the nervous or immune systems, such as diabetes, rheumatoid arthritis, autoimmune diseases, etc.
* Recent Use of Systemic Immunosuppressants: Patients who have recently used systemic immunosuppressive agents.
* Poor Compliance: Patients who are unable to follow up on time or adhere to the treatment plan.
* Pregnancy or Lactation: Pregnant or nursing women, as their physiological state may affect study outcomes.
* Allergy History: Patients with a history of allergies to the study medication or related components.
* Other Reasons: Patients deemed by the investigator to have other reasons making them unsuitable for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Neovascularization Area | 1、2、4、8、12 week
Corneal Clarity Score | 1、2、4、8、12 week
Best Corrected Visual Acuity (BCVA) | 1、2、4、8、12 week
Conjunctival Hyperemia Score | 1、2、4、8、12 week
Corneal Endothelial Cell Count | 1、2、4、8、12 week

CONTACTS AND LOCATIONS:
Locations (1):
- 1 Xihu Avenue, Shangcheng District,Hangzhou, Zhejiang,China,Hangzhou, Zhejiang Completed, Hangzhou, Zhejiang, China